CLINICAL TRIAL: NCT01019863
Title: Study to Evaluate an Oxaliplatin-based Chemotherapy in Patients With Resistant or Relapsing Non-Hodgkin Lymphoma.
Acronym: LNH-RGDOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Dr Rami Kotb, hematologist, CHUS Hopital Fleurimont
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122752
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2009-11

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin (Experimental): oxaliplatin associated with Rituxan,Gemcitabine, and Dexamethasone in patients with refractory or relapsed Non hodgkinien lymphoma
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin — oxaliplatin 100mg/m2 + Rituxan 375 mg/m2 + Gemcitabine 1000mg/m2 every 2 weeks for 8 cycles

SUMMARY:
Evaluation of the efficacy, tolerance, quality of life and cost effectiveness of the association of Oxaliplatin, Gemcitabine, Rituximab and Dexamethasone for treatment of patients with refractory or relapsing non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or above at the time of inclusion.
2. Documented CD20+ NHL, refractory or relapsing after first line chemotherapy.
3. No contraindication to Oxaliplatin, Gemcitabine, Dexamethasone or Rituximab.

Exclusion Criteria:

1. Other types of non-Hodgkin lymphoma
2. Pregnancy and lactation.
3. Patient unable to give written informed consent.
4. Contra-indication ou intolerance to any of the components of the RGDOx chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Response rate to RGDOx in patients with relapsing or refractory NHL | Within 3 months after chemotherapy (6-8 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Kotb, MD, Principal Investigator — CHUS Hopital Fleurimont
Locations (2):
- Canada (2):
  - CHA Hôpital de l'Enfant-Jésus, Québec, Quebec
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec